CLINICAL TRIAL: NCT00791557
Title: An Open Label Single Center Pilot Study Investigating the Clinical Response and Mechanism of Action of Infliximab in the Treatment of Adults With Inflammatory Bowel Disease Who Have Moderate to Severe Pyoderma Gangrenosum
Brief Title: Open Label Study for Adults With Pyoderma Gangrenosum and Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Principal Investigator, Neil Korman, Principle Investigator, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-07-14
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-09

CONDITIONS: Pyoderma Gangrenosum; Crohn's Disease; Ulcerative Colitis; Inflammatory Bowel Disease
MeSH Terms: conditions — Pyoderma Gangrenosum; Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infliximab (Experimental): Single arm open label IV Infliximab given at weeks 1,2,14,22
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — IV drug given at weeks 1,2,14,22
  Other Names: Remicade

SUMMARY:
Subjects must be 18- 75 years old and have a history of both inflammatory bowels disease (Crohn's or ulcerative colitis) and pyoderma gangrenosum.

This is a 6 month open label study of an intravenous (IV) medication. Visits occur every 2 weeks initially, then every 1-2 months later in the study.

ELIGIBILITY:
Inclusion Criteria:

* Must Be ages 18-75
* Must have both inflammatory bowel disease and moderate to severe pyoderma gangrenosum
* Must never have received Infliximab for the treatment of pyoderma gangrenosum

Exclusion Criteria:

* Have had any previous treatment with monoclonal antibodies other than infliximab used to treat IBD or antibody fragments.
* Have a history of serious infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil J Korman, MD.PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab: Single arm open label
  Infliximab : IV drug given at weeks 1,2,14,22
Period: Overall Study
Arm/Group | Infliximab
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab
Number analyzed (Participants) | 2
Age, Customized [Number; unit: participants]
  <=18 years | 0
  Between 18 and 75 years | 2
  >=75 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: The Efficacy of Infliximab in Pyoderma Gangrenosum in Adult Subjects Who Have Inflammatory Bowel Disease
Description: Outcome was measured by clinical assessment of pyoderma gangrenosum. The number of patients who had improvement and/or clearance of the pyoderma grangrenosum after the infusions and through the follow up visit was assessed.
Time Frame: Week 26
Population: Subjects who completed all required transfusions of infliximab were analyzed.
Measure: Number; unit: participants
Arm/Group | Infliximab
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Arm/Group | Infliximab
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=2)
Infusion reaction (Blood and lymphatic system disorders) | 1 (1)
Bone marrow suppression (Blood and lymphatic system disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to timing of the study, only 2 subjects were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes